CLINICAL TRIAL: NCT02828488
Title: Analysis of the Impact of the Fragility of the Over 70 Years of TIA (Transient Ischemic Attack) Prognosis
Brief Title: Analysis of the Impact of the Fragility of the Over 70 Years of TIAprognosis
Acronym: AIT70
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: AIT70
Record Dates: First submitted 2016-07-07; First posted 2016-07-11 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Vascular; Stoke; Ischemic; Transient Ischemic Attack
MeSH Terms: conditions — Ischemia; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — It is a descriptive study. No intervention

SUMMARY:
Fragility, geriatric concept recent identification is defined by simple physical indicators. The literature suggests that it is related to the risk of hospitalization, falls, institutionalization and death. Some studies have shown a link with heart disease, including heart failure. The link with the TIA (transient ischemic attack) has however never been studied. A fortiori, the impact of the fragility of the risk of recurrent stroke after TIA is unknown.

Several questions need to be asked: Among older patients hospitalized for TIA, what proportion of those completing the criteria of frailty? In this same population, is there a correlation between fragility and scores ABCD2 score itself predictive of the risk of subsequent ischemic stroke? In other words, fragile subjects who have a TIA Have a higher risk of ischemic stroke (which could cause a strengthening of prevention measures)?

DETAILED DESCRIPTION:
Hypotheses :

* Frailty is common among the elderly patient population who have a TIA. Compared to control groups of literature.
* Patients with high fragility score ABCD2 also have a high score.
* Patients with a high score of fragility also have a significant number of vascular risk factors (including atrial fibrillation)
* Patients with a high score of fragility also have an average length of stay (ALOS) higher than the others. So underlying the question is: can we learn to better identify patients who are going to need a bigger structure their output at home.

objectives:

* Assess the feasibility of placing a fragile test in acute phase of AIT in USINV.
* To evaluate the frequency of frailty among the population of elderly patients who have a TIA.
* Compare in AIT over 70 years those with fragile high score to those with low scores, especially for ABCD2 score, vascular risk factors and the DMS.
* Statements parameters:

  o The fragility score:
* Choice of fragility score: among the fragility of scores, the most used in international literature is the score of Linda Fried. Moreover, the stress of the study is related to the environment of the USINV (shortly, short DMS, often tired patients). It is therefore important to use this study for a test only, but quick handover. The score Fried also has the advantage (J Gerontol A Biol Sci Med Sci 2001, 56 (3): M146-56) The first 4 items are simple clinical evaluation. The 5th (grip test) will be performed with a device (single gauge measuring the fingers bending strength) loan from the geriatric ward.

ELIGIBILITY:
Inclusion Criteria:

* The TIA is defined pragmatically: any sudden deficit with blood systematization ≤ 1 hour. Among these "TIA", we know that a subgroup may possibly have an MRI with diffusion lesion, indicating a recent ischemic stroke. This subgroup of transient accident is recognized as being at higher risk of recurrence. This criterion will be taken into account in the data analysis.

Exclusion Criteria:

* history of stroke with Rankin score of ≥ 2.
* Dementia
* Severe depression
* evolutionary Cancer
* Heart Failure

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All TIA patients over 70 years hospitalized ICU neurovascular at GHPSJ (Groupe Hospitalier Paris Saint Joseph):
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2015-08-06 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Fried Score for fragility | Day 1

SECONDARY OUTCOMES:
ABCD Score | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: BRUANDET Marie, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No